CLINICAL TRIAL: NCT02860039
Title: Comparison of High vs. Standard Dose Flu Vaccine in Pediatric Stem Cell Transplant Recipients
Brief Title: High Dose Flu Vaccine in Treating Children Who Have Undergone Donor Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Natasha Halasa, MD, Professor of Pediatrics, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VICC PED 1647; NCI-2016-01090 (Registry Identifier: Clinical Trial Reporting Program)
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Results first posted 2022-04-14 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Hematopoietic Cell Transplantation Recipient; Malignant Neoplasm; Influenza
MeSH Terms: conditions — Neoplasms; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - High Dose TIV (Experimental): Patients receive HD-TIV intramuscularly (IM) on day 0 and day 28.
  Interventions: Biological: Trivalent Influenza Vaccine; Other: Laboratory Biomarker Analysis
- Group 2 - Standard Dose QIV (Active Comparator): Patients receive standard dose QIV IM on day 0 and day 28.
  Interventions: Biological: Quadrivalent Influenza Vaccine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Trivalent Influenza Vaccine — High dose Trivalent Influenza Vaccine given intramuscular
  Arms: Group 1 - High Dose TIV
Biological: Quadrivalent Influenza Vaccine — Standard dose Quadrivalent Influenza Vaccine given intramuscular
  Arms: Group 2 - Standard Dose QIV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II randomized trial studies how well high dose flu vaccine works in treating children who have undergone done stem cell transplant. Higher dose flu vaccine may build a better immune response and may provide better protection against the flu than the standard vaccine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether high-dose trivalent inactivated influenza vaccine (HD-TIV) compared with standard dose quadrivalent inactivated influenza vaccine (QIV) will increase the probability of achieving a >= 4-fold rise in hemagglutination-inhibition (HAI) titers, >= 1:40 HAI titer, or higher geometric mean titer (GMT) to influenza A antigens in pediatric hematopoietic stem cell transplant (HSCT) recipients.

SECONDARY OBJECTIVES:

I. To determine whether HD-TIV compared with standard dose QIV will increase the probability of achieving a >= 4-fold rise in HAI titers, >= 1:40 HAI titer, or higher GMT titers to influenza B antigens in pediatric HSCT recipients.

II. To determine the frequency and severity of solicited local injection site adverse events (e.g. pain/ tenderness, redness, and swelling at injection site) with HD-TIV compared to standard QIV in pediatric HSCT recipients.

III. To determine the frequency and severity of solicited systemic adverse events (e.g. fevers, headache, fatigue/malaise, nausea, body ache/myalgia, general activity level, and vomiting) with HD-TIV compared to standard dose QIV in pediatric HSCT recipients.

IV. To define the relationship between HAI titers, in vivo T and B cell phenotype, and in vitro influenza-specific T and B cell response in pediatric HSCT recipients receiving either HD-TIV or standard dose QIV.

V. To correlate HAI responses to microneutralization responses.

VI. To compare the persistent HAI and microneutralization (MN) titers for all four antigen seven months after the last vaccine dose to assess for persistence of antibody titers.

VII. To compare influenza detection by PCR during influenza season in pediatric HSCT recipients receiving either HD-TIV or standard dose QIV.

VIII. To assess HAI and MN response in children vaccinated during year 1 and revaccinated during year 2 using the same antigen dose.

OUTLINE: Patients are randomized to 1 of 2 treatment groups.

GROUP I (Experimental): Patients receive HD-TIV intramuscularly (IM) on day 0 and day 28.

GROUP II (Standard): Patients receive standard dose QIV IM on day 0 and day 28.

After completion of study treatment, patients are followed up at 28-42 days, and at 7 months.

ELIGIBILITY:
1. Inclusion criteria

   1. Allogeneic HSCT recipients who are 3-35 months post-transplant;
   2. 3-17 years of age, inclusive;
   3. Available for duration of study;
   4. Patients with stable GVHD for at least 4 weeks will be eligible (stable is defined as having no major increases in systemic immunosuppressive therapy for GVHD; adjustments of established medications to obtain a stable target level are acceptable and do not impact eligibility). Parent/legal guardian willing and capable of signing written informed consent;
   5. Parent/legal guardian expected to be available for entire study;
   6. Parent/legal guardian can be reached by telephone and/or electronic communication.
   7. Subjects must have a platelet count of ≥30,000 to receive the immunizations. Patients requiring platelet transfusions are eligible to enroll and must have a platelet count ≥30,000 within 72 hours prior to their immunization, or platelet count ≥75,000 without transfusion documented within 30 days for subjects <12 months post-transplant and within 90 days for subjects 12-35 months post-transplant.
2. Exclusion criteria

   1. History of hypersensitivity to previous influenza vaccination or severe hypersensitivity to eggs/egg protein;
   2. History of Guillain-Barre syndrome;
   3. Evidence of hematologic malignancy or disease relapse post-transplant (stable mixed chimerism is permitted);
   4. History of receiving current year seasonal influenza vaccine post-transplant;
   5. Pregnant female;
   6. History of proven influenza disease after September 1, 2018 prior to enrollment
   7. Non-allogeneic (e.g. autologous) or syngeneic hematopoietic SCT recipients;
   8. History of known active infection with HIV, Hepatitis B or Hepatitis C;
   9. History of known severe latex hypersensitivity;
   10. Subjects who have received stem cell boost or delayed donor lymphocyte infusion within 90 days prior to enrollment, including day of enrollment;
   11. Receipt of IVIG/SCIG <27 days prior to calendar day of vaccination;
   12. Subjects who have participated in year 1 and/or 2 of the study, and received study vaccine

Criteria for temporarily delaying vaccine administration: The following conditions are temporary or self-limiting, and a subject may be included in the study once the condition has resolved, provided that the subject is otherwise eligible: 1). Fever ≥100.4ºF/38.0ºC (oral measurement), or an acute illness within 48 hours of enrollment 2). Receipt of any live vaccines within four weeks or any inactivated vaccines within two weeks prior to potential study vaccination.

Note: if patients were eligible for vaccine 1, they will be eligible to receive vaccine 2 regardless of any changes on their GVHD status, unless it is deemed not medically safe to receive influenza vaccine.

For subjects who were enrolled and vaccinated in 2016-17, 2017-18, or 2018-19, the goal is to enroll individuals who participated in the previous influenza season year and administer the same vaccination as the previous year. These subjects are referred to as repeaters. For example, subjects enrolled in 2016-17 could re-enroll in 2017-18, subjects enrolled in 2017-18 could re-enroll in 2018-19, and subjects in 2018-19 are deemed eligible to re-enroll in 2019-20 as repeaters. Subjects may only enroll as a repeater one time and must enroll the year after their original enrollment. Subjects must receive at least one vaccine to be eligible as a repeater in the subsequent year.

Enrollment Criteria for Subjects who Participated in the previous influenza season

* Repeaters will retain their original study ID and their randomization number
* Previous screen failures will not be enrolled.
* If visit 4 from the previous influenza season and visit 1 from the current influenza season year occur on the same day, lab results from visit 4 (prior to consent) can be part of visit 1.

  1. Inclusion criteria

     1. Available for duration of study;
     2. Patients with stable GVHD for at least 4 weeks will be eligible (stable is defined as no major change in systemic immunosuppressive therapy for worsening GVHD; adjustment of actual dose to obtain a stable target level is acceptable).
     3. Subjects must have a platelet count of ≥30,000 to receive the immunizations. Patients requiring platelet transfusions are eligible to enroll and must have a platelet count ≥30,000 within 72 hours prior to their immunization, or platelet count ≥75,000 without transfusion documented within 30 days for subjects <12 months post-transplant and within 90 days for subjects 12-35 months post-transplant.
     4. Parent/legal guardian willing and capable of signing written informed consent;
     5. Parent/legal guardian expected to be available for entire study;
     6. Parent/legal guardian can be reached by telephone and/or electronic communication.
  2. Exclusion criteria

     1. History of hypersensitivity to previous influenza vaccination or severe hypersensitivity to eggs/egg protein;
     2. History of Guillain-Barre syndrome;
     3. Evidence of hematologic malignancy or disease relapse post-transplant (stable mixed chimerism is permitted);
     4. History of receiving current year seasonal influenza vaccine post-transplant;
     5. Pregnant female;
     6. History of proven influenza disease after September 1, 2019 but prior to enrollment
     7. History of known active infection with HIV, Hepatitis B or Hepatitis C;
     8. Subjects who have received stem cell boost or delayed donor lymphocyte infusion within 90 days of enrollment, including day of enrollment
     9. Receipt of IVIG/SCIG <27 days prior to calendar day of vaccination
     10. Non-allogeneic (e.g. autologous) or syngeneic hematopoietic SCT recipients;
     11. Subjects who have participated in year 1 and/or 2 of the study and received study vaccine.

Criteria for temporarily delaying vaccine administration: The following conditions are temporary or self-limiting, and a subject may be included in the study once the condition has resolved, provided that the subject is otherwise eligible: 1). Fever ≥100.4ºF/38.0ºC (oral measurement), or an acute illness within 48 hours of enrollment 2). Receipt of any live vaccines within four weeks or any inactivated vaccines within two weeks prior to potential study vaccination.

Note: if patients were eligible for vaccine 1, they will be eligible to receive vaccine 2 regardless of any changes on their GVHD status, unless it is deemed not medically safe to receive influenza vaccine.

Note: Previous Screen failures who were not vaccinated can be enrolled and will be assigned the same study ID number.

Criteria for temporarily delaying vaccine administration: The following conditions are temporary or self-limiting, and a subject may be included in the study once the condition has resolved, provided that the subject is otherwise eligible: 1). Fever ≥100.4ºF/38.0ºC (oral measurement), or an acute illness within 48 hours of enrollment 2). Receipt of any live vaccines within four weeks or any inactivated vaccines within two weeks of study vaccination.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Halasa, MD, MPH, Principal Investigator — Vanderbilt University
Locations (9):
- United States (9):
  - UCSF Children's Hospital, San Francisco, California
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital Research Institute, Seattle, Washington

REFERENCES:
- [Derived] Bahakel H, Spieker AJ, Hayek H, Schuster JE, Hamdan L, Dulek DE, Kitko CL, Stopczynski T, Batarseh E, Haddadin Z, Stewart LS, Stahl A, Potter M, Rahman H, Amarin J, Kalams SA, Bocchini CE, Moulton EA, Coffin SE, Ardura MI, Wattier RL, Maron G, Grimley M, Paulsen G, Harrison CJ, Freedman J, Carpenter PA, Englund JA, Munoz FM, Danziger-Isakov L, Halasa N; Pediatric HCT Flu Study. Immunogenicity and Reactogenicity of High- or Standard-Dose Influenza Vaccine in a Second Consecutive Influenza Season. J Infect Dis. 2025 Feb 4;231(1):e123-e131. doi: 10.1093/infdis/jiae454. PMID 39279435
- [Derived] Schuster JE, Hamdan L, Dulek DE, Kitko CL, Batarseh E, Haddadin Z, Stewart LS, Stahl A, Potter M, Rahman H, Kalams SA, Bocchini CE, Moulton EA, Coffin SE, Ardura MI, Wattier RL, Maron G, Grimley M, Paulsen G, Harrison CJ, Freedman JL, Carpenter PA, Englund JA, Munoz FM, Danziger-Isakov L, Spieker AJ, Halasa NB; Pediatric HCT Flu Study. The Durability of Antibody Responses of Two Doses of High-Dose Relative to Two Doses of Standard-Dose Inactivated Influenza Vaccine in Pediatric Hematopoietic Cell Transplant Recipients: A Multi-Center Randomized Controlled Trial. Clin Infect Dis. 2024 Jan 25;78(1):217-226. doi: 10.1093/cid/ciad534. PMID 37800415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 200 children were targeted with the expectation of a 20% drop out rate, as described in Section C17 in the protocol. We were able to enroll 170 subjects with an 8% dropout rate between Visit 1 and Visit 4.
Period: Overall Study
Arm/Group | Group 1 - High Dose TIV | Group 2 - Standard Dose QIV
Started | 85 | 85
Visit 1 (Study vaccine administered.) | 85 | 85
Visit 2 (Study vaccine administered.) | 84 | 83
Visit 3 | 78 | 83
Visit 4 | 74 | 81
Visit 1 Repeat (This visit was attended by subjects who enrolled for a second year following their first year of enrollment, and the study vaccine was administered. See protocol for criteria.) | 32 | 34
Visit 2 Repeat (This visit was attended by subjects who enrolled for a second year following their first year of enrollment, and the study vaccine was administered. See protocol for criteria.) | 31 | 34
Visit 3 Repeat (This visit was attended by subjects who enrolled for a second year following their first year of enrollment. See protocol for criteria.) | 30 | 34
Visit 4 Repeat (This visit was attended by subjects who enrolled for a second year following their first year of enrollment. See protocol for criteria.) | 26 | 22
Completed (This includes subjects who completed all four visits for their first year of enrollment. This does not account for those who participated in a "repeater" year.) | 74 | 81
Not Completed | 11 | 4
Not completed — Death | 4 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not otherwise eligible | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of their assigned vaccine
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - High Dose TIV | Group 2 - Standard Dose QIV | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 85 | 85 | 170
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 11.7811 [7.0775 to 14.2508] | 10.6476 [7.0173 to 14.2235] | 10.8694 [7.0173 to 14.2508]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 36 | 76
  Male | 45 | 49 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 17 | 36
  Not Hispanic or Latino | 66 | 68 | 134
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 12 | 31
  White | 55 | 62 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: Immunogenicity as Measured by the Number of Subjects Who Achieve a 4-fold (or Greater) Rise in Post-vaccination HAI Titers
Description: Point estimates and 95% confidence intervals for proportion of subjects achieving seroconversion (4-fold or greater rise in HAI titers from visit 1).
Time Frame: Visit 1 (baseline) was day 0; visit 2 was 28-42 days after visit 1; visit 3 was 28-42 days after visit 2; and visit 4 was 138-222 days after visit 2.
Population: The number analyzed for each row represents the number of participants that completed the indicated visit and had a recorded HAI titer for the indicated antigen and visit.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group 1 - High Dose TIV | Group 2 - Standard Dose QIV
Number analyzed (Participants) | 85 | 85
proportion of participants
  A/H1N1 Visit 2: number analyzed (Participants) | 83 | 83
  A/H1N1 Visit 2 | 0.20 [0.13 to 0.30] | 0.20 [0.13 to 0.30]
  A/H1N1 Visit 3: number analyzed (Participants) | 76 | 80
  A/H1N1 Visit 3 | 0.42 [0.31 to 0.53] | 0.31 [0.22 to 0.42]
  A/H1N1 Visit 4: number analyzed (Participants) | 70 | 76
  A/H1N1 Visit 4 | 0.31 [0.21 to 0.43] | 0.29 [0.20 to 0.40]
  A/H3N2 Visit 2: number analyzed (Participants) | 83 | 83
  A/H3N2 Visit 2 | 0.22 [0.14 to 0.31] | 0.14 [0.08 to 0.23]
  A/H3N2 Visit 3: number analyzed (Participants) | 76 | 80
  A/H3N2 Visit 3 | 0.41 [0.30 to 0.52] | 0.31 [0.22 to 0.42]
  A/H3N2 Visit 4: number analyzed (Participants) | 70 | 77
  A/H3N2 Visit 4 | 0.36 [0.25 to 0.47] | 0.35 [0.25 to 0.46]
  B/Victoria Visit 2: number analyzed (Participants) | 83 | 82
  B/Victoria Visit 2 | 0.24 [0.16 to 0.34] | 0.23 [0.15 to 0.33]
  B/Victoria Visit 3: number analyzed (Participants) | 76 | 79
  B/Victoria Visit 3 | 0.46 [0.35 to 0.57] | 0.46 [0.35 to 0.57]
  B/Victoria Visit 4: number analyzed (Participants) | 70 | 77
  B/Victoria Visit 4 | 0.34 [0.24 to 0.46] | 0.38 [0.28 to 0.49]
  B/Yamagata Visit 2: number analyzed (Participants) | 83 | 83
  B/Yamagata Visit 2 | 0.12 [0.06 to 0.20] | 0.25 [0.17 to 0.35]
  B/Yamagata Visit 3: number analyzed (Participants) | 76 | 80
  B/Yamagata Visit 3 | 0.20 [0.12 to 0.30] | 0.41 [0.31 to 0.52]
  B/Yamagata Visit 4: number analyzed (Participants) | 70 | 77
  B/Yamagata Visit 4 | 0.19 [0.11 to 0.29] | 0.42 [0.31 to 0.53]

2. Secondary Outcome: Proportion of Solicited Local and Systemic Adverse Events
Description: The proportion of subjects in each group experiencing at least one solicited AE with 95% posterior credible intervals, separated by vaccine number and adverse event type. AEs were assessed by clinicians using Tables 4 and 5 within section C16 of the protocol.
  Solicited injection site AEs included: pain, tenderness, erythema/redness, and swelling/induration. The diameter of any erythema/redness and swelling/induration was measured to evaluate "redness size" and "swelling size." Solicited systemic AEs included: fevers, fatigue/malaise, headache, nausea, body ache/myalgia, generally activity, and vomiting.
Time Frame: Up to 7 days following each vaccination: up to day 7 for vaccine 1 and up to day 35-49 for vaccine 2
Population: The number of subjects analyzed for Vaccine 1 represents the number of subjects who attended Visit 1 and received the first vaccine. The number of subjects analyzed for Vaccine 2 represents the number of subjects who attended Visit 2 and received the second vaccine.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group 1 - High Dose TIV | Group 2 - Standard Dose QIV
Number analyzed (Participants) | 85 | 85
proportion of participants
  Vaccine 1 - Fever | 0.024 [0.003 to 0.082] | 0.012 [0.000 to 0.064]
  Vaccine 1 - Fatigue | 0.188 [0.112 to 0.288] | 0.235 [0.150 to 0.340]
  Vaccine 1 - Headache | 0.165 [0.093 to 0.261] | 0.153 [0.084 to 0.247]
  Vaccine 1 - Nausea | 0.129 [0.066 to 0.220] | 0.141 [0.075 to 0.234]
  Vaccine 1 - Myalgia | 0.188 [0.112 to 0.288] | 0.153 [0.084 to 0.247]
  Vaccine 1 - General activity | 0.129 [0.066 to 0.220] | 0.188 [0.112 to 0.288]
  Vaccine 1 - Vomiting | 0.071 [0.026 to 0.147] | 0.071 [0.026 to 0.147]
  Vaccine 1 - Pain | 0.341 [0.242 to 0.452] | 0.341 [0.242 to 0.452]
  Vaccine 1 - Tenderness | 0.435 [0.328 to 0.547] | 0.424 [0.317 to 0.536]
  Vaccine 1 - Redness size | 0.035 [0.007 to 0.100] | 0.035 [0.007 to 0.100]
  Vaccine 1 - Swelling | 0.106 [0.050 to 0.192] | 0.082 [0.034 to 0.162]
  Vaccine 1 - Swelling size | 0.047 [0.013 to 0.116] | 0.024 [0.003 to 0.082]
  Vaccine 2 - Fever: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Fever | 0.071 [0.027 to 0.149] | 0.072 [0.0270 to 0.151]
  Vaccine 2 - Fatigue: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Fatigue | 0.179 [0.104 to 0.277] | 0.1181 [0.105 to 0.280]
  Vaccine 2 - Headache: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Headache | 0.143 [0.076 to 0.236] | 0.157 [0.086 to 0.253]
  Vaccine 2 - Nausea: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Nausea | 0.131 [0.067 to 0.222] | 0.133 [0.068 to 0.225]
  Vaccine 2 - Myalgia: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Myalgia | 0.060 [0.020 to 0.133] | 0.157 [0.086 to 0.253]
  Vaccine 2 - General activity: number analyzed (Participants) | 84 | 83
  Vaccine 2 - General activity | 0.107 [0.050 to 0.194] | 0.169 [0.095 to 0.267]
  Vaccine 2 - Vomiting: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Vomiting | 0.048 [0.013 to 0.117] | 0.048 [0.013 to 0.119]
  Vaccine 2 - Pain: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Pain | 0.345 [0.245 to 0.457] | 0.253 [0.164 to 0.360]
  Vaccine 2 - Tenderness: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Tenderness | 0.429 [0.321 to 0.541] | 0.265 [0.174 to 0.373]
  Vaccine 2 - Redness size: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Redness size | 0.083 [0.034 to 0.164] | 0.048 [0.013 to 0.119]
  Vaccine 2 - Swelling: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Swelling | 0.167 [0.094 to 0.264] | 0.072 [0.027 to 0.151]
  Vaccine 2 - Swelling size: number analyzed (Participants) | 84 | 83
  Vaccine 2 - Swelling size | 0.060 [0.020 to 0.133] | 0.048 [0.013 to 0.119]

3. Secondary Outcome: T and B Cell Phenotype Assessed by Mass Cytometry
Description: T and B cell response was assessed at visit 1,visit 2, visit 3, and visit 4.
  Results are incomplete due to pending grant funding for laboratory testing. This outcome will be updated once the funding has been obtained and results are available.
Time Frame: as for outcome 1
Reporting Status: Not Posted, anticipated posting 2024-12

4. Secondary Outcome: T and B Cell Response Assessed by Mass Cytometry and In-vitro Functionality Assays
Description: T and B cell response was assessed at visit 1, an optional visit 5-10 days after visit 1, visit 2, an optional visit 5-10 days after visit 2, visit 3, and visit 4.
  Results are pending due to pending grant funding for laboratory testing. This outcome will be updated once the funding has been obtained and results are available.
Time Frame: Visit 1 (baseline) was day 0; optional visit 1 was 5-10 days after visit 1; visit 2 was 28-42 days after visit 1; optional visit 2 was 5-10 days after visit 2; visit 3 was 28-42 days after visit 2; and visit 4 was 138-222 days after visit 2.
Reporting Status: Not Posted, anticipated posting 2024-12

5. Secondary Outcome: Percentage of Individuals in Each Group Who Test Positive for Influenza
Description: The percentage of breakthrough flu in vaccinated participants, separated by treatment group.
Time Frame: During the influenza season, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - High Dose TIV | Group 2 - Standard Dose QIV
Number analyzed (Participants) | 85 | 85
Participants | 11 | 13

ADVERSE EVENTS:
Time Frame: AEs and SAEs will be collected through 7 days following each vaccination (up to day 7 for vaccine 1 and up to day 35-49 for vaccine 2). Adverse events will be followed until resolution or until considered stable.
Arm/Group | Group 1 - High Dose TIV | Group 2 - Standard Dose QIV
All-Cause Mortality (participants affected / at risk) | 4/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 17/85 | 9/85
Other Adverse Events (participants affected / at risk) | 1/85 | 2/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - High Dose TIV (N=85) | Group 2 - Standard Dose QIV (N=85)
Viral illness (Infections and infestations) | 4 (5) | 0 (0)
Group A Streptococcus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Metapneumovirus (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
RSV (Infections and infestations) | 2 (2) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Coronavirus (Infections and infestations) | 0 (0) | 1 (1)
Influenza B and RSV (Infections and infestations) | 1 (1) | 0 (0)
C. difficile/Salmonella (Infections and infestations) | 1 (1) | 0 (0)
BK Virus (Infections and infestations) | 0 (0) | 1 (1)
Pansinusitis (Infections and infestations) | 0 (0) | 1 (1)
Allergic contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI GVHD (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 1 (1)
Opioid withdrawal (General disorders) | 0 (0) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Adenovirus (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - High Dose TIV (N=85) | Group 2 - Standard Dose QIV (N=85)
Fever (General disorders) | 0 (0) | 2 (2)
Swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02860039/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT02860039/SAP_001.pdf
  • Informed Consent Form (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02860039/ICF_002.pdf